CLINICAL TRIAL: NCT00058097
Title: Phase II Study of R115777 for the Treatment of Adults With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Tipifarnib and Radiation Therapy in Treating Patients With Newly Diagnosed Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03013; NABTT 2200; CDR285732; U01CA062475 (NIH)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — tipifarnib; Radiotherapy; Radiation

ARMS (1):
- Treatment (tipifarnib) (Experimental): INDUCTION THERAPY: Patients receive oral tipifarnib twice daily for 3 weeks. Treatment repeats every 4 weeks for up to 3 courses.
  RADIOTHERAPY: Within 14 days after the completion of induction therapy, patients undergo radiotherapy daily, 5 days a week, for 6 weeks.
  MAINTENANCE THERAPY: Two weeks after the completion of radiotherapy, patients receive additional tipifarnib as in induction therapy.
  Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: tipifarnib; Radiation: radiation therapy

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation

SUMMARY:
Phase II trial to study the effectiveness of combining tipifarnib with radiation therapy in treating patients who have newly diagnosed glioblastoma multiforme. Tipifarnib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining tipifarnib with radiation therapy may make the tumor cells more sensitive to radiation therapy and may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate overall survival in newly diagnosed patients with glioblastoma multiforme treated with R115777 before (and possibly after) radiation therapy.

SECONDARY OBJECTIVES:

I. To estimate response rate in adult patients with newly diagnosed glioblastoma multiforme treated with R115777 prior to therapy with radiation.

II. To estimate progression free survival in newly diagnosed patients with glioblastoma multiforme treated with R115777 before (and possibly after) radiation therapy.

III. To describe the toxicity associated with this regimen in adult patients with newly diagnosed glioblastoma multiforme.

OUTLINE: This is a multicenter study.

INDUCTION THERAPY: Patients receive oral tipifarnib twice daily for 3 weeks. Treatment repeats every 4 weeks for up to 3 courses.

RADIOTHERAPY: Within 14 days after the completion of induction therapy, patients undergo radiotherapy daily, 5 days a week, for 6 weeks.

MAINTENANCE THERAPY: Two weeks after the completion of radiotherapy, patients receive additional tipifarnib as in induction therapy.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 2 months.

PROJECTED ACCRUAL: A minimum of 54 patients will be accrued for this study within 11-14 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed supratentorial grade IV astrocytoma (glioblastoma multiforme)
* Patients must not have received prior radiation therapy, chemotherapy, hormonal therapy, immunotherapy or therapy with biologic agents (including immunotoxins immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy) or hormonal therapy for their brain tumor; glucocorticoid therapy is allowed
* Patients must have measurable and contrast-enhancing tumor on the post operative, pretreatment MRI/CT scan (within two weeks of starting treatment)
* Patients must have recovered from the immediate post-operative period and be maintained on a stable corticosteroid regimen from the time of their baseline scan until the start of treatment
* Patients must have a Karnofsky performance status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others)
* Absolute neutrophil count >= 1500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dl
* Creatinine =< 1.5 mg/dl
* Total bilirubin =< 2.0 mg/dl
* Transaminases =< 4 times above the upper limits of the institutional norm
* Patients must be able to provide written informed consent and must be aware of the investigational nature of this study
* Patients with the potential for pregnancy or impregnating their partner must agree to follow acceptable birth control methods to avoid conception; the anti-proliferative activity of this experimental drug may be harmful to the developing fetus or nursing infant; female patients of child-bearing potential must have a negative pregnancy test
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix and breast; patients with prior malignancies must be disease-free for >= five years
* Patients must have a mini-mental state exam score (MMSE) of >= 15

Exclusion Criteria:

* Patients with serious concurrent infection or medical illness which would jeopardize the ability of the patient to receive the chemotherapy outlined in this protocol with reasonable safety
* Patients who are pregnant or breast-feeding
* Patients who have received prior radiation therapy, chemotherapy, hormonal therapy (except glucocorticoids), immunotherapy or therapy with biologic agents (including immunotoxins, immunoconjugates, antisense, peptide receptor antagonists, interferons, interleukins, TIL, LAK or gene therapy) for their brain tumor
* Patients receiving concurrent investigational agents
* Patients who have received Gliadel wafer therapy may not participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2003-08; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years
  95% confidence intervals will be estimated.

SECONDARY OUTCOMES:
Response rate | Up to 5 years
  Estimated with 95% confidence intervals.
Progression free survival | Up to 5 years
  Estimated with 95% confidence intervals.
Toxicities, graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) v4.0 | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lustig, Principal Investigator — New Approaches to Brain Tumor Therapy Consortium
Locations (1):
- New Approaches to Brain Tumor Therapy Consortium, Baltimore, Maryland, United States